CLINICAL TRIAL: NCT01103544
Title: Usage of Vinflunine i.v. (JAVLOR®) for the Treatment of Advanced or Metastatic Transitional Cell Carcinoma of the Urothelium in Adult Patients After Failure of a Cisplatinum-containing Therapy
Brief Title: JAVLOR® Online Non-Interventional Trial
Acronym: JONAS-1
Status: Completed | Type: Observational
Sponsor: Pierre Fabre Pharma GmbH (Industry)
Collaborators: DocCheck Medical Services GmbH (Unknown)
Responsible Party: Sponsor
Other Study IDs: JONAS-1
Record Dates: First submitted 2010-04-11; First posted 2010-04-14 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Transitional Cell Carcinoma
Keywords: TCCU; advanced TCCU; metastatic TCCU; transitional cell carcinoma of the urothelium; advanced transitional cell carcinoma of the urothelium; metastatic transitional cell carcinoma of the urothelium; Cisplatinum failure; Vinflunine; Javlor; daily routine; concomitant antiemetic treatment; concomitant antiobstipative treatment; concomitant antiobstipative diet; patient compliance; quality of life; non-interventional study; Germany; Advanced / metastatic TCCU after Cisplatinum-failure
MeSH Terms: conditions — Carcinoma, Transitional Cell; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with advanced / metastatic TCCU after CDDP-failure

SUMMARY:
Documentation of data concerning tolerability and efficacy of the intravenous treatment with vinflunine performed under daily routine conditions in Germany. The trial focusses on tolerability including the assessment of the usage of anti-emetic and anti-obstipative concomitant treatment as well as on the efficacy of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Legally competent male and female patients
* Advanced or metastatic transitional cell carcinoma of the urothelium
* Failure of a prior Cisplatinum-containing treatment
* Performance Status 0 or 1
* Signed patient informed consent

Exclusion Criteria:

* Missing signed patient informed consent
* Performance Status 2 or higher
* Life expectancy < 2 months
* Brain metastases
* Creatinine-clearance < 20 ml/min
* Child-Pugh-stadium C
* Prothrombin time < 50%
* Bilirubin > 5 x ULN
* Transaminases > 6 x ULN
* Gamma-Glutamyl-transferase > 15 x ULN
* Pregnant or breast-feeding women
* Known/suspected hypersensitivity against vinflunine or other vinca-alkaloids
* Recent (within the last 2 weeks) or current severe infections
* Baseline ANC < 1,500/mm3 or platelets < 100,000/mm3
* Patients being institutionalised due to court/regulatory order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced or metastatic transitional cell carcinoma of the urothelium after failure of a Cisplatinum-containing therapy
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-09 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Side effects according to NCI-CTCAE v3.0 and treatment conditions in daily routine | 9 months after LPI

SECONDARY OUTCOMES:
Explorative assessment of Overall Response Rate (ORR) | 9 months after LPI
Anti-emetic comedication | 9 months after LPI
Anti-obstipative diet / comedication | 9 months after LPI
General well-being / quality of life of the patients (patient questionnaire) | 9 months after LPI
Patients' satisfaction with the treatment (patient questionnaire) | 9 months after LPI
Physicians' satisfaction with the treatment | 9 months after LPI
Patients' compliance with regards to the cotreatments (patient questionnaire) | 9 months after LPI

CONTACTS AND LOCATIONS:
Locations (1):
- Pierre Fabre Pharma GmbH, Freiburg im Breisgau, Germany